CLINICAL TRIAL: NCT03139656
Title: Assessment of the Predictors and Moderators of Health Behavior Change
Acronym: ABC3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Michael Otto, Investigator, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4345E
Record Dates: First submitted 2017-04-28; First posted 2017-05-04 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Health Behaviors
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Values Clarification (Experimental): This intervention will incorporate elements from several widely established self-regulatory strategies aimed at enhancing the motivational aspects of goal pursuit, including mental contrasting (Oettingen, 2000), self-reflection (Koestner et al., 2002), self-affirmation (Schmeichel and Vohs, 2009), and the values clarification components of Acceptance and Commitment Therapy (ACT; Hayes, Strosahl, & Wilson, 1999). Participants will be prompted to enter their selected health goal and will then be instructed to identify personal values that might be practiced in pursuit of this goal. Participants will write about these values for several minutes, after which they will be instructed to select a short phrase or image that conjures up for them the reasons they choose to engage in their goal. Participants will be asked to type the phrase into a textbox and will have the option of receiving a confidential print-out of their chosen phrase at the end of the study visit.
  Interventions: Behavioral: Values Clarification
- Planning (Experimental): Participants in this condition will be guided to create detailed implementation intentions, or if-then planning statements (Gollwitzer & Sheeran, 2006), specifying when, how, and where they will engage in their selected health goal. Participants will be provided with a detailed rationale adapted from earlier research on implementation intentions (e.g., Webb et al., 2010). Participants will be guided to generate a plan indicating when, where, and how they will enact their goal-based behavior over the next week. They will also be prompted to identify 3 obstacles they are likely to encounter during the pursuit of each goal, and to specify in an "if-then" format what specific actions they will take to overcome each obstacle (following the procedures and sample "if-then" responses of Koestner et al., 2002). They will be asked to rehearse each "if-then" statement to themselves before the end of the visit.
  Interventions: Behavioral: Planning
- Combined (Values Clarification & Planning) (Experimental): Participants in this condition will complete abbreviated versions of both the "values clarification" and "planning" procedures, as detailed above. Participants will be prompted to identify 2 obstacles (as opposed to 3) they might encounter during the pursuit of each goal. For each of the obstacles they identify with respect to each of their target goals, they will be prompted to form an additional implementation intention in the form: "When [I encounter the specified obstacle], I will do [X] and remember [values-based statement or image identified during "values clarification" exercise]." They will be asked to rehearse these "if-then" statements to themselves before the end of the visit.
  Interventions: Behavioral: Combined

INTERVENTIONS:
Behavioral: Values Clarification — This intervention will incorporate elements from several widely established self-regulatory strategies aimed at enhancing the motivational aspects of goal pursuit, including mental contrasting (Oettingen, 2000), self-reflection (Koestner et al., 2002), self-affirmation (Schmeichel and Vohs, 2009), and the values clarification components of Acceptance and Commitment Therapy (ACT; Hayes, Strosahl, & Wilson, 1999). Participants will be prompted to enter their selected health goal and will then be instructed to identify personal values that might be practiced in pursuit of this goal. Participants will write about these values for several minutes, after which they will be instructed to select a short phrase or image that conjures up for them the reasons they choose to engage in their goal. Participants will be asked to type the phrase into a textbox and will have the option of receiving a confidential print-out of their chosen phrase at the end of the study visit.
  Arms: Values Clarification
Behavioral: Planning — Participants in this condition will be guided to create detailed implementation intentions, or if-then planning statements (Gollwitzer & Sheeran, 2006), specifying when, how, and where they will engage in their selected health goal. Participants will be provided with a detailed rationale adapted from earlier research on implementation intentions (e.g., Webb et al., 2010). Participants will be guided to generate a plan indicating when, where, and how they will enact their goal-based behavior over the next week. They will also be prompted to identify 3 obstacles they are likely to encounter during the pursuit of each goal, and to specify in an "if-then" format what specific actions they will take to overcome each obstacle (following the procedures and sample "if-then" responses of Koestner et al., 2002). They will be asked to rehearse each "if-then" statement to themselves before the end of the visit.
  Arms: Planning
Behavioral: Combined — Participants in this condition will complete abbreviated versions of both the "values clarification" and "planning" procedures, as detailed above. Participants will be prompted to identify 2 obstacles (as opposed to 3) they might encounter during the pursuit of each goal. For each of the obstacles they identify with respect to each of their target goals, they will be prompted to form an additional implementation intention in the form: "When [I encounter the specified obstacle], I will do [X] and remember [values-based statement or image identified during "values clarification" exercise]. They will be asked to rehearse these "if-then" statements to themselves before the end of the visit.
  Arms: Combined (Values Clarification & Planning)

SUMMARY:
This study will investigate three interventions-values clarification, planning, or combined (values clarification + planning)-for increasing goal-consistent health behavior (e.g., exercise or dieting). The investigators will also examine how intervention effects differ based on various psychological and neuropsychological factors, to better understand how interventions can be tailored to specific individuals.

The investigators hypothesize a) that the combined intervention will increase goal-consistent exercise behavior more than the other interventions; and b) that individuals scoring higher on self-concordance or goal-commitment will benefit more from planning, whereas those with more positive expectancies or scoring higher on neuropsychological measures (e.g., working memory) will benefit more from values clarification.

DETAILED DESCRIPTION:
The study will be a repeated measures design examining the between-subjects effect of intervention condition (values clarification, planning, and combined) on self-reported health goal progress and related outcomes at 1-week and 4-week follow-up, relative to baseline. Based on this design, participants will first be instructed to generate a health-related goal on which they want to make progress over the course of the next month (following procedures adapted from Little, 1993, and Sheldon & Kasser, 1998; see details below). Participants will then be randomly assigned (using a random number table) to one of three intervention conditions: (1) values clarification, (2) planning, and (3) combined (values clarification + planning). All conditions are described in more detail below. Fifty-three participants will be randomized to each condition. Questionnaire measures assessing a variety of psychological variables as well as neuropsychological measures will be modeled as between-subject predictor and/or moderator variables of goal-consistent health behavior. Additionally, differences in self-concordance, goal commitment, and expectancies of success will be modeled as potential moderator and/or mediator variables.

ELIGIBILITY:
Inclusion Criteria:

* Boston University Psychology 101 students at least 18 years of age
* Able to provide informed consent for the study
* Sufficient command of the English language
* Have experience using a computer and mouse

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Goal Progress | Change from baseline to 1-week and 4-week follow-ups
  This 3-item goal progress measure assesses participants' self-reported effort towards and success at meeting their specified goal over the past week, each on a 7-point Likert scale. The third item assesses the number of actions participants have undertaken to realize their goal in the past week (previously shown to be a valid indicator of goal pursuit; Oettingen et al., 2001; Sevincer & Oettingen, 2009).

SECONDARY OUTCOMES:
Perceived Locus of Causality (PLOC) | Change from baseline to 1-week and 4-week follow-ups
  The PLOC scale (Sheldon & Kasser, 1995, 1998) is a 4-item measure of the level of autonomy or self-concordance that participants experience with respect to a given goal.
Positive and Negative Affect Schedule (PANAS) | Change from baseline to 1-week and 4-week follow-ups
  Participants rate 20 adjectives describing positive and negative affect states on a 5-point Likert scale indicating to what extent they currently feel that way.
Goal Rating Measure | Change from baseline to 1-week and 4-week follow-ups
  On a 7-point Likert scale, participants will rate their health-related goal regarding their expectancies of success, their energization towards the goal, and the perceived difficult and importance of the goal.
Goal Orientation Scale | Change from baseline to 1-week and 4-week follow-ups
  This is a 5-item scale that assesses participant's orientation toward a growth/learning-focused versus fixed/performance-focused motivation, adapted from Brett and VandeWalle (1999).
Action Control Scale - Preoccupation subscale | Change from baseline to 1-week and 4-week follow-ups
  This is an abbreviated version of the scale designed by Diefendorff et al. (2000).
Distress Intolerance Index (DII) | Change from baseline to 1-week and 4-week follow-ups
  The DII is a 10-item self-report questionnaire consisting of items from four commonly used distress intolerance measures.
Penn State Worry Questionnaire--Brief Version | Change from baseline to 1-week and 4-week follow-ups
  The Brief Penn State Worry Questionnaire (Brief PSWQ;Topper et al., 2014) is a 5-item self-report scale that assess the tendency to worry.
Self-Control Scale | Change from baseline to 1-week and 4-week follow-ups
  The SCS (Tangney et al., 2004) is a 10-item measure of ability to implement self-control across varying situations.
Delay Discounting Task | Change from baseline to 1-week and 4-week follow-ups
  The Delay Discounting Task adapted from Kirby and Marakovic (1996) evaluates the degree to which participants are willing to delay rewards.
Need for Cognition Scale (Short Form) | Change from baseline to 1-week and 4-week follow-ups
  The NCS-SF (Cacioppo, Petty, & Kao, 1984) is an 18-item scale that assesses the characteristic tendency to enjoy and seek out cognitively challenging tasks and activities.
Cognitive Reflection Test (CRT) | Change from baseline to 1-week and 4-week follow-ups
  The CRT (Frederick, 2005) is a 3-item task that assesses the tendency to use "fast," intuitive heuristic-based reasoning versus "slow," more deliberative reasoning
Implicit Attitudes toward Effort | Change from baseline to 1-week and 4-week follow-ups
  The investigators will use an adapted version of the Brief Implicit Association Test (B-IAT; Sriram & Greenwald, 1998) to assess participants' implicit tendency to appraise the experience of effort as either "good" or "bad."
Satisfaction with Life Scale (SWLS) | Change from baseline to 1-week and 4-week follow-ups
  The SWLS (Diner, Emmons, Larsen, & Griffin, 1985) is a 5-item scale assessing global cognitive judgments of one's current life satisfaction.
Center for Epidemiological Studies Depression Scale (CES-D) | Change from baseline to 1-week and 4-week follow-ups
  The CES-D (Radloff, 1977) is a 20-item measure of items relating to or indicating symptoms of depression experienced over the past week.
Beck Anxiety Inventory (BAI) | Change from baseline to 1-week and 4-week follow-ups
  The BAI (Beck, Epstein, Brown, & Steer, 1988) is a commonly used 21-item, self-report inventory designed to measure severity of anxiety symptoms.
Generalized Self-Efficacy Scale (GSE) | Change from baseline to 1-week and 4-week follow-ups
  The GSE (Schwarzer & Jerusalem, 1995) is a 10-item scale designed to assess optimistic self-beliefs used to cope with a variety of demands in life.
Ruminative Responses Scale--Brief Version | Change from baseline to 1-week and 4-week follow-ups
  The Brief Ruminative Responses Scale (Brief RRS; Topper et al., 2014) is a 5-item self-report scale that assess the tendency to ruminate.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No